CLINICAL TRIAL: NCT06907459
Title: Effect of Release of Upper Track of Deep Front Facial Line Versus Myofascial Release With IASTM on Patients With Upper Cross Syndrome
Acronym: UCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator : alshaymaa shaaban abd el azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005666
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Upper Cross Syndrome
Keywords: upper cross syndrome; IASTM; Release of Upper Track of Deep Front Facial Line
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: release upper track of frontal line facia and IASTM
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper Track of Deep Front Facial Line realese (Experimental): Thirty subjects received release of upper track of deep front facial line in addition supervised corrective exercises three times a week for four weeks.
  Interventions: Other: upper Track of Deep Front Facial Line realese; Other: supervised corrective exercises
- Myofascial Release With IASTM (Experimental): thirty subjects received myofascial release with IASTM in addition supervised corrective exercises three time a week for four weeks
  Interventions: Other: Myofascial Release With IASTM; Other: supervised corrective exercises
- supervised corrective exercises (Active Comparator): thirty subjects received supervised corrective exercises three time a week for four weeks
  Interventions: Other: supervised corrective exercises

INTERVENTIONS:
Other: upper Track of Deep Front Facial Line realese — The MFR techniques were applied to the designated regions, with soft, steady pressure lasting 90 to 120 seconds postural correction exercises The upper track of deep front facial line release procedures were applied. Hyoid mobilization; Larynx mobilization; Sternal oscillations; and Barral's Transversus Thoracis mobilization. The thoracic inlet releasing ; intrathoracic fascia elongation; scalene releasing and diaphragm relaxation
  Arms: Upper Track of Deep Front Facial Line realese
Other: Myofascial Release With IASTM — The instrument is designed to mobilize soft tissues. Facilitation approaches were employed to break apart adhesions. Emollient Gel/Lubrication Gel (Hawk Grips product) was also used to lubricate the skin and allow the instrument to move more easily. The tool has two sides: one for therapy and the other for holding plus postural correction exercises
  Arms: Myofascial Release With IASTM
Other: supervised corrective exercises — The exercise program included cervical stabilization exercises performed in 3 sets of 10 repetitions with a 10-second maintenance, scapular stabilization exercises plus stretching of cervical muscles.

SUMMARY:
this study will be conducted to compare the effect of release of upper track of deep front facial line versus myofascial release with IASTM on patients with Upper Cross Syndrome.

DETAILED DESCRIPTION:
Upper cross syndrome is a postural dysfunction that can cause a variety of upper-body musculoskeletal problems. Early detection and physiotherapy can help to prevent further complications. Maintaining bad posture over an extended duration can cause postural dysfunction and misalignment.

The first and most obvious sign of upper crossed syndrome is the characteristic postural dysfunction of protracted scapulae, medially rotated humeri, hyperkyphotic upper thoracic spine, and a protracted/ anteriorly held head, which is created by hypo lordosis or even kyphosis (excessive flexion) of the lower cervical spine, hyper lordosis of the upper cervical spine and head, and anterior translation of the head upon the atlas.

The available treatments for upper cross syndrome are Stretching, strengthening, myofascial release, postural relaxation exercise, electrical stimulations, and deep neck flexors activations are the most used techniques. Numerous studies have highlighted various benefits in terms of time efforts, and prognosis. Those are corrective exercise, Kinesio taping, scapular stabilization exercise, and PNF techniques.

Studies have demonstrated the role of fascia in various musculoskeletal dysfunctions as the fascial tissues connect the skeletal muscles forming a body-wide web in a pattern called myofascial meridians. As fascia is able to modify its tensional state, strain transmission along the meridians might occur in response to changes in muscle activity.

Deep fascia tends to be highly vascularized and contain well developed lymphatic channels. In some instances, deep fascia can even contain free encapsulated nerve endings, such as Ruffini and Pacinian corpuscles. It is present in our body in different tissue planes and in different forms with specific function and the musculoskeletal fascial system can be affected by various localized disorders with variable time course and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years old
* All participants had forward head, craniovertebral angle < 50.
* All participants had rounded back (kyphosis angle ≥ 42°)
* Based on assessment of upper cross syndrome by photogrammetric analysis.
* The subjects were chosen from both genders.

Exclusion Criteria:

* History of trauma or surgery in cervical region.
* Bone fractures or acute soft tissue injuries.
* Osteoporosis.
* Heart attack.
* Unstable angina pectoris -Implanted pacemaker or defibrillator- -Cancer-
* Rheumatoid arthritis
* Connective tissue disease: This includes diseases such as osteomyelitis, lupus and scleroderma -Neurological conditions-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
neck disability | up to four weeks
  The neck disability assessment will be performed using the Neck Disability Index (NDI) questionnaire - it contains ten items that refer to neck pain (intensity) and the level of ability to manage daily living activities (personal care, reading, lifting, headache, work, concentration, driving, sleep and recreation). The NDI score is interpreted as 0-4=no disability, 5-14=mild disability, 15-24=moderate disability, 25-34=severe disability, and over 34= total disability, where a score of 50 converted to percentiles represents 100%. NDI score is calculated as follows: total score/total possible score, transformed to percentage multiplied by 100=% points

SECONDARY OUTCOMES:
pain intensity | up to four weeks
  he subject was in a relaxed position then gave him the appendix which contains VAS. The subject was instructed to place a vertical mark on the line to indicate his/her pain. the line has two ends; one with no pain (zero) and the other extreme pain (100 mm) at the other end
craniovertebral angle | up to four weeks
  craniovertebral angle will be measured by Photogrammetry method. A CVA below 48-50 degrees indicates FHP
kyphosis angle | up to four weeks
  kyphosis angle will be measured by Photogrammetry method.
upper chest expansion | up to four weeks
  tape measurements will be used to measure upper chest expansion
lower chest expansion | up to four weeks
  ape measurements will be used to measure lower chest expansion
cervical range of motion | up to four weeks
  cervical range of motion device will be used to measure cervical range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Alshaymaa Shaaban Abdelazeim, Giza, Dokki, Egypt